CLINICAL TRIAL: NCT06731504
Title: A Pilot Trial of Abatacept Based Graft-Versus-Host Disease Prophylaxis Following Omidubicel Hematopoietic Cell Transplantation
Brief Title: HMCT/CT2401: Abatacept GVHD Prophylaxis Following Omidubicel HCT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00116015
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Abatacept/tacrolimus/mycophenolate mofetil (ABA/Tac/MMF) following omidubicel HCT (Experimental): Abatacept 10 mg/kg is given on day -1, +5, +14, and +28 in combination with standard of care tacrolimus and mycophenolate mofetil-based GVHD prophylaxis. This regimen will follow an omidubicel transplantation.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Abatacept is a monoclonal antibody that suppresses T-cell activation through costimulatory blockade. In 2021, abatacept was FDA approved to prevent acute GVHD following allogeneic HCT.

SUMMARY:
This study is a single-center, non-randomized, single-arm pilot trial of omidubicel hematopoietic stem cell transplantation (HCT) for hematologic malignancies with myeloablative conditioning chemotherapy of physician's choice followed by abatacept/tacrolimus/mycophenolate mofetil (ABA/Tac/MMF) graft-versus-host disease (GVHD) prophylaxis. The primary objective is to assess the safety and feasibility of abatacept/tacrolimus/mycophenolate mofetil GVHD prophylaxis following omidubicel HCT.

Target enrollment is 10 participants. Subjects are adults with a diagnosis of hematologic malignancy with an available cord blood unit for omidubicel product manufacturing. Patients will be followed for a total of 18 months and will have research blood draws and Abatacept pharmacokinetics, as well as standard of care assessments that will be reviewed for this study.

It is estimated that 36 months of accrual will be necessary to enroll the targeted sample size with an accrual rate of approximately 1 participant every 3 months. Accrual will be reported by race, ethnicity, gender, and age. Descriptive analyses are planned given the sample size.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of hematologic malignancy with an available cord blood unit for omidubicel product manufacturing
2. Adult patients (≥18 at the time of enrollment)
3. Adequate organ function for transplant defined as:

   1. Left ventricular ejection fraction ≥ 40%;
   2. DLCO, FEV1, FVC > 50% predicted;
   3. Total bilirubin ≤ 2.5 mg/dL except for patients with Gilbert's syndrome or hemolysis, and ALT, AST, and alkaline phosphatase all < 5 x upper limit of normal (ULN);
   4. Serum creatinine within normal range, or if serum creatinine outside normal range, must have measured or estimated creatinine clearance > 40 mL/min/1.73m2;
   5. Karnofsky performance score ≥ 70; and
   6. If applicable, > 6 months since a previous autologous transplant.
4. Female patients (unless postmenopausal or surgically sterilized) and male patients (even if surgically sterilized) must agree to practice two effective methods of contraception at the same time, or agree to completely abstain from heterosexual intercourse from the time of signing informed consent through 100 days post-transplant. Fertility preservation method will be left to treating physician's discretion.

Exclusion Criteria:

1. Patients with known sensitivity to dimethyl sulfoxide, dextran 40, gentamicin, human serum albumin or bovine material
2. Presence of a donor-specific antibodies with MFI >2000
3. Uncontrolled bacterial, fungal or viral infection
4. Treatment with any other investigational medical product (medications without any known FDA approved indication) needs to be discussed with the PI for patient eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Safety of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as evaluated by frequency of adverse events. | 6 months post-HCT
  Adverse events are defined by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. Only events related to Abatacept (and not solely expected toxicities of omidubicel HCT) will be recorded.
Safety of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as evaluated by severity of adverse events. | 6 months post-HCT
  Adverse events are defined by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. Only events related to Abatacept (and not solely expected toxicities of omidubicel HCT) will be recorded.
Feasibility of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as evaluated by number of subjects who receive minimum dose of ABA. | Day 28 post-HCT
  Minimum dose is 4 doses of minimum 10mg/kg of abatacept prophylaxis following omidubicel transplant.

SECONDARY OUTCOMES:
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by Severe GVHD-Free and Progression-Free Survival (SRFS). | 18 months post-HCT
  Severe GVHD-Free and Progression-Free Survival (SRFS) as a time to event outcome is defined as the first event of Grade III-IV acute GVHD or chronic GVHD requiring systemic immune suppression, with underlying disease progression or relapse, and death by any cause.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by rates of acute GVHD. | 18 months post-HCT
  Cumulative incidences of Grade II-IV and III-IV acute GVHD will be determined per Glucksberg criteria.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by rates of chronic GVHD - mild, moderate, and severe per NIH criteria. | 18 months post-HCT
  The cumulative incidence of chronic GVHD will be determined per NIH Consensus Conference Criteria.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by hematologic recovery. | 30 days post-HCT
  Hematologic recovery is defined by achieving both neutrophil and platelet count recovery after transplant. Neutrophil recovery is defined as achieving an absolute neutrophil count (ANC) greater than or equal to 500/mm3 for three consecutive measurements on three different days. Platelet recovery is defined as the first day of a sustained platelet count (1) greater than or equal to 20,000/mm3 or (2) greater than or equal to 50,000/mm3 with no platelet transfusions in the preceding seven days.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by rates of severe infections at 6 months post-transplant. | 6 months post-HCT
  The incidence of definite and probable viral, fungal, and bacterial infections will be tabulated.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by rates of viral reactivations at 6 months post-transplant. | 6 months post-HCT
  The cumulative incidence of treated CMV and HHV6 reactivation in the first 6 months post-transplant will be described.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by donor cell engraftment. | Day 28, 60, and 90 post-HCT
  Donor cell engraftment will be assessed by donor/recipient chimerism studies. Chimerism may be evaluated in bone marrow, whole unfractionated blood, or blood cell fractions, including CD3 and CD33 or CD15 fraction.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by disease relapse or progression. | Day 90 post-HCT
  Relapse or progression will be diagnosed by bone marrow assessment.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by non-relapse mortality (NRM). | Day 100, 180, and 365 post-HCT
  NRM is defined as death without evidence of disease progression or recurrence.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by disease-free survival (DFS). | 18 months post-HCT
  DFS is defined as the time from date of transplant to death or relapse/progression, whichever comes first.
Efficacy of ABA/Tac/MMF GVHD prophylaxis following omidubicel HCT as measured by overall survival (OS). | 18 months post-HCT
  OS is defined as the time interval between date of transplant and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Sanghee Hong, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No